CLINICAL TRIAL: NCT04769557
Title: Pre-emptive Analgesics for Additional Pain Relief in Impacted Third Molar Surgery by depositing4% Articaine With 1:200000 Epinephrine Using Vazirani-Akinosi Closed Mouth Technique- A Randomized Clinical Trial
Brief Title: Pre Emptive Analgesics for Pain Relief in Impacted Lower Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Abdul Kalam Azad, Assistant Professor, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MMMC/FOD/AR/B5/E C-2017(07)
Record Dates: First submitted 2021-02-06; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Experimental): Paracetamol
  Interventions: Drug: paracetamol
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paracetamol — tablet paracetamol 500 mg
  Other Names: Paracetamol 500 mg
  Arms: Paracetamol
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of pre-emptive paracetamol in reducing intra operative pressure and post operative pain after surgical removal of impacted mandibular third molar using visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years and above
* Healthy patients (ASA I)
* Patients who are not allergic to the drugs and local anesthetic agents used

Exclusion Criteria:

* Patients who are on concurrent treatment with NSAIDs or corticosteroids
* Patients with pericoronitis or periapical infection

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
intraoperative pain | during luxation of tooth
  A 10 mm Visual Analogue Scale with higher score depicting severe pain
postoperative pain | 1 day
  A 10 mm Visual analogue scale with higher score depicting severe pain

SECONDARY OUTCOMES:
Time to rescue medication | upto 360 minutes
  minutes
number of patients taking rescue medications | Upto 360 minutes
  Total number of patients taking rescue medications

CONTACTS AND LOCATIONS:
Overall Officials: Abdul K azad, MDS, Principal Investigator — Melaka Manipal Medical College
Locations (1):
- Melaka manipal medical college, Malacca, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP